CLINICAL TRIAL: NCT03481062
Title: Optimisation of Subclavian Venous Catheterization
Brief Title: Anatomy and Ultrasound Evaluation for Central Venous Access
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OSCAR
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Catheterization, Central Venous; Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Neutral
- abduction
- pad
- combination

SUMMARY:
The anatomy and ultrasound image of subclavian vein was investigated on cadavers, volunteers and patients, respectively. Structures，approach，position and complications were discussed to improve the success rate and safety of central venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* gender unlimited
* 18.5 < body mass index (BMI) < 30
* written consent signed.

Exclusion Criteria:

* abnormality of the infraclavicular region, including infection, deformity,
* history of bone, joint, muscle or neurovascular disease
* history of injury, radiation or invasive procedure
* subjects refused.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult Asian without past medical history of the infraclavicular region
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
area | 12 months
  SV area in square centimeter
length | 12 months
  SV length in centimeter

SECONDARY OUTCOMES:
width | 12 months
  SV width in centimeter
skin distance | 12 months
  depth from skin in centimeter
comfort | 12 months
  comfort level rated by Likert scale ranged point 1 to 5, indicating increased comfort level

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China